CLINICAL TRIAL: NCT01556477
Title: A Multicentre Open Randomized Phase II Study of the Efficacy and Safety of Azacitidine Alone or in Combination With Lenalidomide in High-risk Myeloid Disease (High-risk Myelodysplastic Syndrome and Acute Myeloid Leukemia) With a Karyotype Including Del(5q)
Brief Title: The Efficacy of Azacitidine +/- Lenalidomide in High-risk Myelodysplastic Syndrome (MDS)and Acute Myeloid Leukemia (AML) With Del(5q).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordic MDS Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMDSG10B; 2011-001639-21 (EudraCT Number)
Record Dates: First submitted 2012-03-12; First posted 2012-03-16 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Myelodysplastic Syndrome; Acute Myelogenous Leukemia
Keywords: MDS; AML; Azacitidine; Lenalidomide; del5q
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azacitidine (Active Comparator)
  Interventions: Drug: Azacitidine
- azacitidine + lenalidomide (Experimental)
  Interventions: Drug: azacitidine + lenalidomide

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 5-2-2 (75 mg/m2/day subcutaneously for 5 days, followed by a 2-day weekend break, followed by azacitidine 75 mg/m2/ day for 2 days every 28 days, no individual dose exceeding 200 mg) for 6 cycles.
  Other Names: Vidaza
  Arms: azacitidine
Drug: azacitidine + lenalidomide — Azacitidine 5-2-2 (75 mg/m2/day subcutaneously for 5 days, followed by a 2-day weekend break, followed by azacitidine 75 mg/m2/ day for 2 days every 28 days, no individual dose exceeding 200 mg) for 6 cycles.
  Initial dose of lenalidomide is 10 mg 21/28 days, starting day 1 in each azacitidine cycle and leaving the last week before start of next azacitidine cycle free. The dose should increased to 25 mg day 1 in cycle 4 if no toxicity according to predefined criteria occurs. Total treatment period is 24 weeks.
  Other Names: Vidaza and Revlimid
  Arms: azacitidine + lenalidomide

SUMMARY:
The proposed phase II trial is a multicenter, randomized, open-label study that will evaluate the efficacy and safety of azacitidine alone or in combination with lenalidomide in high-risk Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML) with a karyotype including del(5q). The primary objective will be to evaluate the efficacy in terms of response according to International Working Group (IWG) criteria for MDS and AML after 6 cycles of azacitidine or azacitidine + lenalidomide treatment, or at end of study if this occurs at an earlier time point.

DETAILED DESCRIPTION:
This is an prospective open multi-center randomized phase II study of standard dose azacytidine with or without the addition of lenalidomide in high-risk myeloid disease (high-risk MDS and AML) with a karyotype including del(5q). Seventy-two patients, eligible for treatment with azacytidine (Intermedium/INT-2 and High-risk MDS and AML with 20-30 % marrow blasts according to label) will be included.

Azacytidine will be given in a modified standard dose, azacytidine 5+2 (75 mg/m2/ d subcutaneously for 5 days, followed by a 2-day weekend break, followed by azacytidine 75 mg/m2/ d for 2 days every 28 days, no individual dose exceeding 200 mg) for 6 cycles. Cycle interval may be prolonged if toxicity according to predefined criteria occurs. Patients will be randomized to azacytidine (Arm A) or azacytidine + lenalidomide (Arm B). The initial dose of lenalidomide is 10 mg 21/28 days, starting day 1 in each azacytidine cycle and leaving the last week before start of next azacytidine cycle free. The dose should be increased to 20 mg day 1 in cycle 4 if no toxicity according to predefined criteria occurs. The total study period is 24 weeks + additional weeks caused by prolonged cycle interval. Patients, who following a response may be eligible for allo-SCT may exit the study after cycle 3, 4 or 5 and then be subject to end-of-study assessment. Patients who at start of treatment, or any time during study have a neutrophil count <0,5 x 109/l will be treated with Granulocyte-ColonyStimulatingFactor (G-CSF).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at the time of signing the informed consent form.
* MDS with IPSS Int-2 or High with a karyotype including del(5q).
* Acute myeloid leukaemia (AML) with multilineage dysplasia and 20-30 % blasts (former RAEB-t) with a karyotype including del(5q).
* Subject has signed the informed consent form.
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test prior to starting lenalidomide. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, patches, or implantable hormonal contraceptive methods; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on lenalidomide. WCBP must agree to have pregnancy tests every 4 weeks while on lenalidomide.
* Males (including those who have had a vasectomy) must use barrier contraception (latex condoms) when engaging in reproductive sexual activity with WCBP while on lenalidomide, when temporarily stopping lenalidomide and 28 days after the last dose of lenalidomide.

Note: Refractory and relapsed patients can be included as long as they fulfil the inclusion criteria.

Exclusion Criteria:

* Eligible for upfront allogeneic SCT without prior induction chemotherapy or azacitidine
* Pregnant or lactating females.
* Prior therapy with azacitidine
* Prior therapy with lenalidomide
* Expected survival less than two months.
* Acute promyelocytic leukemia (APL)
* Central nervous system leukemia
* Serum biochemical values as follows

  1. Serum creatinine >2.0 mg/dL (177 mmol/L)
  2. Serum aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transferase (ALT)/serum glutamate pyruvate transaminase (SGPT) >3.0 x upper limit of normal (ULN)
  3. Serum total bilirubin >1.5 mg/dL
* Prior allergic reaction to thalidomide
* Uncontrolled systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-07 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Response according to IWG criteria for MDS and AML | 25-44 weeks (after 6 cycles of azacitidine or azacitidine+lenalidomide)
  Response according to IWG criteria include hematologic response (including transfusion independence), bone marrow response (blast count) and cytogenetic response (karyotype) after 6 cycles of azacytidine or azacytidine+lenalidomide. For patients who can keep the 4 week interval the Time Frame will be 25 weeks. The cycle interval can be extended up to 8 weeks which makes 44 weeks the maximum Time Frame.

SECONDARY OUTCOMES:
Cytogenetic response after 3 cycles using Fluorescence In Situ Hybridization(FISH) | 25-44 weeks
  After 3 cycles the 5q- clone will be measured with FISH to see if there is a response already at that time. For patients who can keep the 4 week interval the Time Frame will be 25 weeks. The cycle interval can be extended up to 8 weeks which makes 44 weeks the maximum Time Frame.
Safety (number and types of adverse advents) in azacitidine vs azacitidine + lenalidomide groups | 25-44 weeks
  Heamtological adverse events will be monitored by checking Hemoglobin,Leucocyte count, Platelet and a Differential every week. Non-Hematological adverse events will be monitored and reported in the Case report form (CRF). For patients who can keep the 4 week interval the Time Frame will be 25 weeks. The cycle interval can be extended up to 8 weeks which makes 44 weeks the maximum Time Frame.
Azacitidine cycle interval between groups | 25-44 weeks
  For patients who can keep the 4 week interval the Time Frame will be 25 weeks. The cycle interval can be extended up to 8 weeks which makes 44 weeks the maximum Time Frame.
Survival in azacitidine vs azacitidine + lenalidomide groups | Up to week 156
  All patients will undergo follow-up once yearly from start of treatment; week 52, 104, and 156.
Relapse in azacitidine vs azacitidine + lenalidomide groups | Up to week 156
  All patients will undergo follow-up once yearly from start of treatment; week 52, 104, and 156.
Analysis of a broad spectrum of molecular and cellular events which previously have been identified as related to MDS with del(5q). | 25-44 weeks
  Bone marrow will be biobanked at inclusion and after 6 cycles of treatment or or at end of study if this occurs at an earlier time point. For patients who can keep the 4 week interval the Time Frame will be 25 weeks. The cycle interval can be extended up to 8 weeks which makes 44 weeks the maximum Time Frame.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Möllgård, MD, PhD, Principal Investigator — Nordic MDS Group
Locations (1):
- Lars Möllgård, Stockholm, Sweden

REFERENCES:
- [Derived] Rasmussen B, Nilsson L, Tobiasson M, Jadersten M, Garelius H, Dybedal I, Gronbaek K, Ejerblad E, Lorenz F, Flogegard M, Marcher CW, Cavalier L, Ebeling F, Olsnes AM, Norgaard JM, Saft L, Mollgard L, Hellstrom-Lindberg E, Schlegelberger B, Gohring G. Influence of Cytogenetics on the Outcome of Patients With High-Risk Myelodysplastic Syndrome Including Deletion 5q Treated With Azacitidine With or Without Lenalidomide. Genes Chromosomes Cancer. 2025 Feb;64(2):e70029. doi: 10.1002/gcc.70029. PMID 39921387
- See also: Nordic MDS Group website — http://www.nmds.org